CLINICAL TRIAL: NCT02728804
Title: Implementation of a Prospective Financial Impact Assessment Tool in Patients With Metastatic Colorectal Cancer
Brief Title: S1417CD Financial Impact Assessment Tool in Patients With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S1417CD; NCI-2015-01885 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1417; S1417CD (Other: SWOG); SWOG-S1417CD (Other: DCP); S1417CD (Other: CTEP); UG1CA189974 (NIH); NCT02755571 (obsolete NCT alias)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Health Services Research (questionnaire administration): Patients complete questionnaires (including the Baseline, Financial/Employment Impact, Insurance Impact, Quality of Life, and Treatment Perceptions questionnaires) over 30-60 minutes at baseline and at 3, 6, 9, and 12 months. Caregivers complete questionnaires over 30-60 minutes at baseline and at 6 and 12 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete questionnaire
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial studies the use of the financial impact assessment tool in patients with colorectal cancer that has spread from the primary site to other places in the body. Gathering information about patients with colorectal cancer over time may help doctors better understand the financial impact of cancer and help patients avoid financial problems during treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the incidence of treatment-related major financial hardship over 12 months, among patients with newly diagnosed metastatic colorectal cancer (mCRC) treated at components and subcomponents of the National Cancer Institute (NCI) Community Oncology Research Program (NCORP).

SECONDARY OBJECTIVES:

I. To describe the association of major financial hardships with mCRC treatment by demographic factors, including age, race, marital status, employment status, and income.

II. To explore whether occurrence of major financial hardship is associated with poorer health-related quality of life over time.

III. To profile the magnitude and timing of treatment-related changes in patients' income, assets, debt, and employment, and to quantify major out-of-pocket expenses during the 12 months following registration.

IV. To explore the extent to which health insurance factors (e.g. high copayments, deductibles, premiums, loss/change of insurance plan) are associated with major financial hardship and treatment non-adherence.

V. To determine feasibility of recruiting primary caregivers and measuring caregiver burden and caregivers' perceptions about cancer treatment costs.

VI. To determine the feasibility of conducting a prospective-multi-site longitudinal cohort study assessing financial outcomes in patients with mCRC undergoing treatment within the NCORP network.

TERTIARY OBJECTIVES:

I. To obtain objective measures of expenses, debt and credit through linkage with individual patient credit reports (TransUnion) at enrollment (baseline) and end of follow up (12 months).

OUTLINE:

Patients complete questionnaires (including the Baseline, Financial/Employment Impact, Insurance Impact, Quality of Life, and Treatment Perceptions questionnaires) over 30-60 minutes at baseline and at 3, 6, 9, and 12 months. Caregivers complete questionnaires over 30-60 minutes at baseline and at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed metastatic colon or rectal cancer (mCRC) (de novo metastatic diagnosis) or metastatic recurrence after prior treatment for stage I-III disease and be </= 120 days after diagnosis at time of registration
* Systemic chemotherapy and/or systemic biologic therapy must be planned to be administered within 30 days after registration or must have been initiated within 60 days prior to registration; patients who are planning palliative or hospice care only (no chemotherapy or biologic therapy) are not eligible
* Registering site must be an NCORP site; it is recommended that patients receive care for the mCRC at the registering site to ensure accessibility of patient records.
* Patients must be able to complete questionnaires in English
* Patients must provide their full name, primary address in the United States (U.S.), birth date and social security number at registration for the purposes of accessing credit report data
* Patients must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed metastatic colon or rectal cancer treated at NCORP sites.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veena Shankaran, Principal Investigator — SWOG Cancer Research Network
Locations (537):
- United States (537):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Reid Health, Richmond, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Ochsner Medical Center West Bank, Gretna, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Ochsner Hematology Oncology North Shore - Slidell (East Region), Slidell, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Nevada Cancer Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Boston Baskin Cancer Center-Bartlett, Bartlett, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Integrity Oncology PLLC-Collierville, Collierville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Sovah Health Martinsville, Martinsville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 380 patients were enrolled between June 2016 and January 2019.
Period: Overall Study
Arm/Group | Health Services Research (Questionnaire Administration)
Started | 380
Eligible and Completed Baseline Questionnaire | 368
Completed | 269
Not Completed | 111
Not completed — Ineligible | 3
Not completed — Did not complete baseline questionnaire | 9
Not completed — Death | 99

BASELINE CHARACTERISTICS:
Population: The analysis population includes the 368 participants that are eligible and completed the baseline questionnaire.
Arm/Group | Health Services Research (Questionnaire Administration)
Number analyzed (Participants) | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 231
  >=65 years | 137
Age, Continuous [Median (Full Range); unit: years] | 60.2 [21.1 to 89.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 228
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 17
  Black | 48
  White | 286
  Other or Unknown | 17
Marital Status [Count of Participants; unit: Participants]
  Married/Partnered | 213
  Divorced or separated | 82
  Widowed | 17
  Never married | 48
  Unknown | 8
Primary Insurance [Count of Participants; unit: Participants]
  Private insurance (employer provided) | 171
  Medicare | 143
  Medicaid | 44
  Other | 3
  Uninsured | 7
Total Household Income [Count of Participants; unit: Participants]
  $0-$25,000 | 114
  $25,001-$50,000 | 94
  $50,001-$75,000 | 54
  $75,001-$100,000 | 31
  $100,001 or more | 65
  Unknown | 10
Education [Count of Participants; unit: Participants]
  High school graduate or less | 143
  Vocational school or some college | 111
  Bachelor degree | 63
  Master, doctorate, or professional degree | 43
  Missing | 8
Homeowner [Count of Participants; unit: Participants]
  Yes | 236
  No | 124
  Unknown | 8
Prediagnosis Employment Status [Count of Participants; unit: Participants]
  Employed (full-time, part-time, self-employed) | 222
  Retired | 93
  On leave of absence from paid employment | 2
  Unemployed | 13
  Temporary or permanent disability | 25
  Other or unknown | 13
Total Assets [Count of Participants; unit: Participants]
  $0-$25,000 | 202
  $25,001-$50,000 | 25
  $50,001-$100,000 | 38
  $100,001-$250,000 | 32
  $250,001-$500,000 | 29
  $500,001 or more | 34
  Unknown | 8
Prior Diagnosis of Stage I-III Colorectal Cancer [Count of Participants; unit: Participants]
  Yes | 93
  No, de novo diagnosis of stage IV | 275
ECOG Performance Score [Count of Participants; unit: Participants] — ECOG performance status scores range from 0 to 3, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  Participants
    0 | 183
    1 | 158
    2 | 22
    3 | 4
    Unknown | 1
Initial Treatment Regimen [Count of Participants; unit: Participants]
  (5-FU or cap) ± bevacizumab | 38
  (FOLFOX or CapOX) ± bevacizumab | 228
  (FOLFIRI or CapIRI) ± bevacizumab | 55
  (FOLFOX, CapOX, FOLFIRI, or CapIRI) + EGFR inhibitor | 15
  Other | 32

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence Rate of Treatment-related Major Financial Hardship
Description: The cumulative incidence estimates of participants experiencing both major financial hardship (MFH) and multiple financial hardships will be reported. This estimate is calculated over a 12 month period; due to participant drop out throughout this period, the calculated cumulative incidence for the participants analyzed at the 12 month mark does not equate to a whole number. A major financial hardship is defined as one or more of the following: debt accumulation of any amount, selling or refinancing home, >= 20% income decline, borrowing money of any amount from family/friends.
Time Frame: Up to 12 months
Population: The analysis population includes only the 302 participants that were evaluable for the primary endpoint - either completed 12-month evaluation or met primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Health Services Research (Questionnaire Administration)
Number analyzed (Participants) | 302
percentage of participants
  Any MFH | 71.3 [65.7 to 76.1]
  New Debt | 57.6 [51.7 to 63.0]
  >=20% Income Decline | 26.6 [21.3 to 32.0]
  Loans from Family and/or Friends | 26.0 [21.5 to 30.7]
  Refinance of Home | 3.4 [1.7 to 5.9]
  Sale of Home | 2.6 [1.3 to 4.7]

2. Secondary Outcome: Association of Age and Cumulative Incidence Rate of Major Financial Hardship
Description: The cumulative incidence estimates of participants experiencing MFH within age groups. This estimate is calculated over a 12 month period; due to participant drop out throughout this period, the calculated cumulative incidence for the participants analyzed at the 12 month mark does not equate to a whole number. This is used to assess whether major financial hardship at one year differs by age (< 65 vs. >= 65). Age is taken at baseline.
Time Frame: Up to 12 months
Population: There were a total of 302 participants analyzed which either completed the 12-month evaluation or met the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- < 65 Years; >=65 Years: This group is comprised of eligible and evaluable participants that are under 65 years of age.
Arm/Group | < 65 Years | >=65 Years
Number analyzed (Participants) | 192 | 110
percentage of participants | 73.7 [66.4 to 79.6] | 68.1 [58.6 to 76.0]
Statistical Analysis 1: Comparison: < 65 Years vs >=65 Years; Test type: Superiority; p = 0.65, Regression, Cox; Covariate adjustment for insurance status, education, and sex; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.66 to 1.29]

3. Secondary Outcome: Association of Race and Cumulative Incidence Rate of Major Financial Hardship
Description: The cumulative incidence estimates of participants experiencing MFH within racial groups. This estimate is calculated over a 12 month period; due to participant drop out throughout this period, the calculated cumulative incidence for the participants analyzed at the 12 month mark does not equate to a whole number. This is used to assess whether major financial hardship at one year differs by race (white vs. non-white).
Time Frame: Up to 12 months
Population: 292 total participants were analyzed which had baseline race information available and either completed the 12-month evaluation or met the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- White: This group is comprised of eligible and evaluable participants that identify as White.
- Non-White: This group is comprised of eligible and evaluable participants that identify as a non-White race.
Arm/Group | White | Non-White
Number analyzed (Participants) | 240 | 52
percentage of participants | 70.3 [64.1 to 75.6] | 73.9 [59.4 to 83.9]
Statistical Analysis 1: Comparison: White vs Non-White; Test type: Superiority; p = 0.70, Regression, Cox; Covariate adjustment for insurance status, education, and sex; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.79 to 1.43]

4. Secondary Outcome: Association of Marital Status and Cumulative Incidence Rate of Major Financial Hardship
Description: The cumulative percentage of participants experiencing MFH within marital status groups. This is used to assess whether major financial hardship at one year differs by age (married vs. unmarried). Marital status is taken at baseline.
Time Frame: Up to 12 months
Population: 295 participants were analyzed who had baseline marital status information available and either completed the 12-month evaluation or met the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Not Married: This group is comprised of eligible and evaluable participants that are neither married nor partnered.
- Married: This group is comprised of eligible and evaluable participants that are either married or partnered.
Arm/Group | Not Married | Married
Number analyzed (Participants) | 116 | 179
percentage of participants | 69.0 [60.5 to 76.1] | 72.2 [64.0 to 78.8]
Statistical Analysis 1: Comparison: Not Married vs Married; Test type: Superiority; p = 0.87, Regression, Cox; Covariate adjustment for insurance status, education, and sex; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.73 to 1.31]

5. Secondary Outcome: Association of Employment Status and Cumulative Incidence Rate of Major Financial Hardship
Description: The cumulative incidence estimates of participants experiencing MFH within different employment status groups. This estimate is calculated over a 12 month period; due to participant drop out throughout this period, the calculated cumulative incidence for the participants analyzed at the 12 month mark does not equate to a whole number. This is used to assess whether major financial hardship at one year differs by pre-diagnosis employment status (any employment vs. unemployed). Employment status is taken at baseline.
Time Frame: Up to 12 months
Population: 295 participants were analyzed that had baseline employment status information available and either completed the 12-month evaluation or met the primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Unemployed: This group is comprised of eligible and evaluable participants that are unemployed.
- Any Employment: This group is comprised of eligible and evaluable participants that are employed by any means. This includes full-time employment, part-time employment, self-employed, and on leave from full-time employment.
Arm/Group | Unemployed | Any Employment
Number analyzed (Participants) | 101 | 194
percentage of participants | 62.9 [53.8 to 70.7] | 76.2 [69.2 to 81.9]
Statistical Analysis 1: Comparison: Unemployed vs Any Employment; Test type: Superiority; p = 0.01, Regression, Cox; Covariate adjustment for insurance status, education, and sex; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.48 to 0.92]

6. Secondary Outcome: Association of Income and Cumulative Incidence Rate of Major Financial Hardship
Description: The cumulative incidence estimates of participants experiencing MFH within income groups. This estimate is calculated over a 12 month period; due to participant drop out throughout this period, the calculated cumulative incidence for the participants analyzed at the 12 month mark does not equate to a whole number. This is used to assess whether major financial hardship at one year differs by household income (<$50,000 vs. >=$50,000 and <$100,000 vs. >=$100,000). Household income is taken at baseline.
Time Frame: Up to 12 months
Population: 294 total participants were analyzed which had baseline household income information available and either completed the 12-month evaluation or met the primary endpoint. The number of participants in the <$50,000 arm and >=$50,000 arm equal the total (294) participants analyzed. Similarly, the number of participants in the <$100,000 arm and >=$100,000 arm equal the total (294) participants analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- <$50,000: This group is comprised of eligible and evaluable participants whose yearly income is less than $50,000.
- >=$50,000: This group is comprised of eligible and evaluable participants whose yearly income is at least $50,000.
- <$100,000: This group is comprised of eligible and evaluable participants whose yearly income is less than $100,000.
- >=$100,000: This group is comprised of eligible and evaluable participants whose yearly income is at least $100,000.
Arm/Group | <$50,000 | >=$50,000 | <$100,000 | >=$100,000
Number analyzed (Participants) | 168 | 126 | 239 | 55
percentage of participants | 72.7 [65.6 to 78.6] | 69.1 [59.3 to 77.1] | 72.9 [67.0 to 77.9] | 64.9 [45.6 to 78.8]
Statistical Analysis 1: Comparison: <$50,000 vs >=$50,000; Test type: Superiority; p = 0.10, Regression, Cox; Covariate adjustment for insurance status, education, and sex; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.95 to 1.87]
Statistical Analysis 2: Comparison: <$100,000 vs >=$100,000; Test type: Superiority; p = 0.002, Regression, Cox; Covariate adjustment for insurance status, education, and sex; Hazard Ratio (HR) = 1.92, 95% CI 2-sided [1.28 to 2.89]

7. Secondary Outcome: Health-related Quality of Life (HRQOL) as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) Version 3.0
Description: The relationship between major financial hardship and HRQOL will be assessed. Landmark analysis will be used to establish major financial hardship as a baseline predictor of HRQOL. In particular, patients will be categorized as having major financial hardship at their 3 month assessment (yes vs. no). Linear regression will then be used to assess whether the 3-month assessment of financial hardship predicts the 6-month HRQOL score. HRQOL at 3 months will be included as an adjustment covariate. The 6-month HRQOL score will be based on the EORTC QLQ-C30 questionnaire transformed into a linear sco
Time Frame: Up to 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Changes in Assets/Income/Wealth
Description: Will be handled using descriptive statistics (e.g. mean, median, proportions). Descriptive statistics will be used to summarize baseline patient characteristics and will compare populations using two-sample means and proportions tests (alpha level 0.05). Caregiver strain index will be scored based on responses (score range 0 to 26). Mean scores will be compared for caregivers of patients reporting vs. not reporting at least one financial hardship.
Time Frame: Baseline to up to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Out-of-pocket Expenses, Defined as Total Out-of-pocket Direct Medical (e.g., Prescriptions, Physician Visits, Deductibles) and Non-medical (Transportation, Meals) Expenses in the 3 Months Prior to Each Study Visit
Description: as for outcome 8
Time Frame: Up to 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Changes in Health Insurance
Description: as for outcome 8
Time Frame: Baseline to up to 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Caregiver Participation
Description: The caregiver component will be considered feasible if the designated caregivers for > 50% of eligible patients complete and submit their baseline and at least one follow-up assessment. Means, medians, and proportions will be used to describe the participating caregiver population. Analyses will be largely descriptive. If caregiver accrual is very poor (< 20%), describing the patient population will be the focus rather than attempting to correlate caregiver and patient responses.
Time Frame: Up to 12 months
Reporting Status: Not Posted

12. Secondary Outcome: Accrual to a Prospective-multi-site Longitudinal Cohort Study
Description: Each of the NCORP components (we anticipate 25 NCORP components) will each need to enroll, on average, about 5 patients per year. Accrual will be assessed at 1.5 years after study activation. If monthly average accrual in quarters 5-6 after study registration is < 50% of projected accrual, efforts will be made to increase accrual over the succeeding 6 month period. If after 2 years, monthly accrual remains < 50% of projected accrual, study revision will be considered. In order to address the potential for selection bias, demographics (age, race, gender, etc.) of the final cohort will be compared
Time Frame: Up to 3 years
Reporting Status: Not Posted

13. Secondary Outcome: Debt and Spending by Credit Report Histories
Description: Credit histories obtained from TransUnion measure the following: non-mortgage amounts past due on credit cards and bankcards; non-mortgage credit card and bankcard balances; bankruptcies, liens, collections or repossessions. Will be handled using descriptive statistics (e.g. mean, median, proportions). Descriptive statistics will be used to summarize baseline patient characteristics and will compare populations using two-sample means and proportions tests (alpha level 0.05). Caregiver strain index will be scored based on responses (score range 0 to 26). Mean scores will be compared.
Time Frame: Up to 12 months
Reporting Status: Not Posted

14. Secondary Outcome: Credit History (TransUnion)
Description: The linkage of SWOG clinical and financial data with credit histories obtained from TransUnion will allow exploration of additional indicators of financial stress, including high balances and past due amounts of credit card and bankcards as well as evidence of bankruptcies, liens, and collections or repossessions in the preceding 36 months (TransUnion Inc. 'Credit Vision' report). This linked database will also provide a more complete picture of patients' pre-diagnosis financial status and post-diagnosis financial hardship. These data will also allow corroboration of self-reports.
Time Frame: Up to 12 months
Reporting Status: Not Posted

15. Secondary Outcome: Financial Stress (Patient, Caregiver, or Bereaved Caregiver)
Description: as for outcome 8
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of study participant - up to 12 months.
Description: Serious adverse events and other (non-serious adverse events) were not assessed for the study. All-cause mortality was assessed for the 380 participants at the start of the study.
Arm/Group | Health Services Research (Questionnaire Administration)
All-Cause Mortality (participants affected / at risk) | 99/380
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02728804/Prot_SAP_ICF_000.pdf